CLINICAL TRIAL: NCT01695980
Title: Laryngeal Mask Airway in Pediatric Adenotonsillectomy
Acronym: LMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Cristina Baldassari M.D., Assistant Professor, Pediatric Otolaryngology, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: version 4 25Jun2012
Record Dates: First submitted 2012-09-24; First posted 2012-09-28 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Sleep Apnea, Obstructive; Tonsillitis
Keywords: adenotonsillectomy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Tonsillitis | interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LMA with modified retractor (Experimental): LMA with modified retractor
  Interventions: Other: LMA with modified retractor
- ETT with non modified retractor (Active Comparator): ETT with non modified retractor
  Interventions: Procedure: ETT with non modified retractor

INTERVENTIONS:
Procedure: ETT with non modified retractor — adenotonsillectomy
  Arms: ETT with non modified retractor
Other: LMA with modified retractor — LMA with modified retractor
  Arms: LMA with modified retractor

SUMMARY:
The study will compare how often the tubing kinks when a LMA (laryngeal mask airway) with modified retractor is used compared to use of an endotracheal tube (ETT) and non modified retractor is used.

DETAILED DESCRIPTION:
The laryngeal mask airway (LMA)is a device used to secure the airway of patients during general anesthesia. This device is routinely used for anesthesia in elective head and neck surgeries, including adenotonsillectomy. In this study, the efficacy of the LMA will be studied as it pertains to operative times and cost.

The child will be randomized into either the LMA group or the ETT group.

ELIGIBILITY:
Inclusion Criteria:

* requiring adenotonsillectomy for Obstructive sleep apnea or chronic tonsillitis between the ages of 2-16

Exclusion Criteria:

* children with BMI >35
* unwillingness to comply with study procedures
* children with craniofacial anomalies/abnormalities which will interfere with mask placement
* children under 2 or over 16

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
To determine the number of participants with adverse events with use of LMA and ETT during adenotonsillectomy. | one year
  Mouth gag equipment is used for the LMA and the ETT. A modified tongue depressor is used with the LMA and a non-modified tongue depressor is used with the ETT. Data will be collected in regards to the rate of kinking/obstruction of the tubing with each type of equipment to determine which option is the best for use in adenotonsillectomy.

SECONDARY OUTCOMES:
To determine total length of procedure and recovery time with use the LMA. | One year
  Does the rate of kinking/obstruction of the tubing cause prolonged procedure time and additional issues for anesthesia and the subsequent recovery of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Baldassari, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Children's Hospital of the King's Daughters, Norfolk, Virginia, United States